CLINICAL TRIAL: NCT00803517
Title: Comparison of Multifocal Electroretinogram Assessment Between Laser Treatment Group and Photodynamic Therapy Group in Chronic Central Serous Chorioretinopathy
Brief Title: Comparison of Multifocal Electroretinogram Assessment in Chronic Central Serous Chorioretinopathy (CSC) Between Laser Treatment Group and Photodynamic Therapy Group in Chronic Central Serous Chorioretinopathy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Samsung Medical Center, Samsung Medical Center
Other Study IDs: 2008-05-030
Record Dates: First submitted 2008-11-12; First posted 2008-12-05 (Estimated); Results first posted 2008-12-05 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-02

CONDITIONS: Central Serous Chorioretinopathy
Keywords: chronic central serous chorioretinopathy; multifocal electroretinogram; central retinal function after treatment in chronic serous chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Photodynamic therapy (PDT)
- Focal laser photocoagulation (focal)

SUMMARY:
This study is a comparison of multifocal electroretinogram assessment between the laser treatment group and the photodynamic therapy group in chronic central serous chorioretinopathy.

DETAILED DESCRIPTION:
1. Laser Group: extrafoveal focal leakage on FAG
2. PDT Group: no definite focal leak on FAG subfoveal or juxtafoveal focal leakage on FAG, or serous retinal pigmentary epithelial detachment involving foveal center

Inclusion criteria

1. Chronic serous chorioretinopathy (over 3 months) when subretinal fluid persisted in the subfoveal region demonstrated by clinical examination and OCT
2. Ability to maintain steady fixation for mfERG
3. Presence of abnormal dilated choroidal vasculature in ICGA
4. Symptom duration over 3 months

Exclusion criteria

1. previous PDT or laser treatment history
2. evidence of Choriinal neovascularization in FAG
3. other chorioretinal disorders that can cause macular exudation such as age-related macular degeneration, pathologic myopia, angioid streaks, trauma, inflammatory diseases, retinal vasculopathies, and hereditary dystrophies

follow-up Visit

1)baseline 2)1month 3)3months 4)6 months

each visit: multifocal electroretinogram, visual acuity, optical coference timography should be measured.

ELIGIBILITY:
Inclusion Criteria:

1. CSC (over 3 months) when subretinal fluid persisted in the subfoveal region demonstrated by clinical examination and OCT
2. Ability to maintain steady fixation for mfERG
3. Presence of abnormal dilated choroidal vasculature in ICGA
4. Symptom duration over 3 months

Exclusion Criteria:

1. Previous PDT or laser treatment history
2. Evidence of CNV in FAG
3. Other chorioretinal disorders that can cause macular exudation such as age-related macular degeneration, pathologic myopia, angioid streaks, trauma, inflammatory diseases, retinal vasculopathies, and hereditary dystrophies

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Laser Group: extrafoveal focal leakage on FAG
  2. photodynamic therapy Group: no definite focal leak on FAG subfoveal or juxtafoveal focal leakage on FAG, or s-RPED involving foveal center
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Se Woong Kang, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photodynamic Therapy | Focal Laser Photocoagulation
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photodynamic Therapy | Focal Laser Photocoagulation | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.35 (6.89) | 44.26 (5.89) | 43.31 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Multifocal Electroretinogram Amplitudes
Description: Amplitude at first annular ring at multifocal electroretinogram RETIscan (Roland Consult, Wiesbaden, Germany) is used for multifocal retinogram.
  The recording protocol was chosen according to the International Society for Clinical Electro-physiology of Vision (ISCEV) guidelines.
Time Frame: baseline, 1 month, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Photodynamic Therapy | Focal Laser Photocoagulation
Number analyzed (Participants) | 12 | 12
microvolts
  baseline | 28.4 (8.6) | 32.2 (10.46)
  1 month | 29.7 (7.2) | 36.1 (13.6)
  3 months | 39.9 (8.7) | 37.6 (10.9)
  6 months | 40.3 (6.7) | 38.6 (12.3)

2. Secondary Outcome: Best Corrected Visual Acuity
Description: Best-corrected visual acuities were obtained with Snellen charts. Snellen's visual acuity was converted logarithm of the minimum angle of resolution (logMAR) for statistical analysis.
Time Frame: baseline, 1 month, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Photodynamic Therapy | Focal Laser Photocoagulation
Number analyzed (Participants) | 12 | 12
logMAR
  baseline | 0.22 (0.17) | 0.15 (0.13)
  1 month | 0.07 (0.02) | 0.08 (0.14)
  3 months | 0.05 (0.02) | 0.04 (0.02)
  6 months | 0.05 (0.02) | 0.04 (0.02)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No